CLINICAL TRIAL: NCT01854892
Title: The RELIEF Study - Researching the Effectiveness of Lumbar Interventions for Enhancing Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Responsible Party: Principal Investigator, James Thomas, Professor, Ohio University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: AT006978
Record Dates: First submitted 2013-05-03; First posted 2013-05-16 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Low Back Pain
Keywords: low back pain; manipulation; laser therapy; osteopathic; chiropractic; mobilization; muscle energy; physical therapy; muscle; spine; adjustment; rehabilitation
MeSH Terms: conditions — Low Back Pain | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Manipulation (Experimental): Spinal manipulation
  Interventions: Other: Manipulation
- Mobilization (Experimental): Spinal mobilization
  Interventions: Other: Mobilization
- Laser Therapy (Experimental): Cold laser therapy
  Interventions: Other: Laser Therapy

INTERVENTIONS:
Other: Manipulation — High velocity short amplitude thrust spinal manipulation applied to the lumbar spine.
  Arms: Manipulation
Other: Mobilization — Static isometric contractions of the lumbar spine to induce spinal mobilization
  Arms: Mobilization
Other: Laser Therapy — Cold laser applied to the paravertebral muscles in the lumbar region
  Arms: Laser Therapy

SUMMARY:
Low back pain (LBP) is one of the most common reasons for seeking medical care and accounts for over 3.7 million physician visits/year in the U.S. alone. Ninety percent of adults will experience low back pain in their lifetime, 50% will experience recurrent LBP, and 10% will develop chronic pain and related disability.

While there is growing evidence for the clinical effectiveness of alternative and complementary therapies to treat low back pain, little is known on the physiologic consequences and effects of these treatments. Further, additional data is needed to understand how these different treatment techniques effect clinical changes in pain and disability. The lack of empirical data hinders acceptance by the wider scientific and health-care communities, and it also limits the development of rational strategies for using alternative and complementary therapies.

ELIGIBILITY:
Inclusion Criteria:

* Report history consistent with chronic low back pain
* Average pain intensity at least mild when assessed with a numerical pain scale
* At least mild disability when assessed with a questionnaire
* Meets criteria for clinical prediction rule

Exclusion Criteria:

* A history of certain neurological, cardiorespiratory, and musculoskeletal disorders
* Have active cancer or be blind
* Report recent use of certain medications and treatments
* Report being pregnant, lactating, or that she anticipates becoming pregnant in the next 3-months
* Have too high body mass or unexplained weight loss
* Have clinical depression
* Have pending litigation related to the low back pain or are receiving any type of disability services
* Current drug or alcohol use that would interfere with adherence to study requirements

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2013-06; Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-05 (Actual)

PRIMARY OUTCOMES:
Change in numerical pain rating score | 48 hours post 3 week intervention
Change in disability score | 48 hours post 3 week intervention
  Roland Morris disability questionnaire

SECONDARY OUTCOMES:
Change in score on PROMIS Pain Behavior Survey | 48 hours post 3 week intervention
  This survey was developed by the NIH to provide reliable and valid measures of pain behavior. We will exam the change in scores on this survey from visit 2 (initial testing session) to visit 8(48 hours post 3 week intervention)
Change in scores on PROMIS pain interference survey | 48 hours post 3 week interventions
  This survey was developed by the NIH to provide reliable and valid measures of pain interference. We will exam the change in scores on this survey from visit 2 (initial testing session) to visit 8(48 hours post 3 week intervention)
Change in scores on PROMIS pain intensity survey | 48 hours post 3 week intervention
  This survey was developed by the NIH to provide reliable and valid measures of pain intensity. We will exam the change in scores on this survey from visit 2 (initial testing session) to visit 8(48 hours post 3 week intervention)
Change in scores on PROMIS physical function survey | 48 hours post 3 week intervention
  This survey was developed by the NIH to provide reliable and valid measures of physical function. We will exam the change in scores on this survey from visit 2 (initial testing session) to visit 8(48 hours post 3 week intervention).

CONTACTS AND LOCATIONS:
Overall Officials: James S Thomas, Ph.D., PT, Principal Investigator — Ohio University; Brian C Clark, Ph.D., Principal Investigator — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States

REFERENCES:
- [Derived] Stamenkovic A, Clark BC, Pidcoe PE, van der Veen SM, France CR, Russ DW, Kinser PA, Thomas JS. Distinguishing chronic low back pain in young adults with mild to moderate pain and disability using trunk compliance. Sci Rep. 2021 Apr 7;11(1):7592. doi: 10.1038/s41598-021-87138-6. PMID 33828171
- [Derived] Thomas JS, Clark BC, Russ DW, France CR, Ploutz-Snyder R, Corcos DM; RELIEF Study Investigators. Effect of Spinal Manipulative and Mobilization Therapies in Young Adults With Mild to Moderate Chronic Low Back Pain: A Randomized Clinical Trial. JAMA Netw Open. 2020 Aug 3;3(8):e2012589. doi: 10.1001/jamanetworkopen.2020.12589. PMID 32756930
- [Derived] Clark BC, Russ DW, Nakazawa M, France CR, Walkowski S, Law TD, Applegate M, Mahato N, Lietkam S, Odenthal J, Corcos D, Hain S, Sindelar B, Ploutz-Snyder RJ, Thomas JS. A randomized control trial to determine the effectiveness and physiological effects of spinal manipulation and spinal mobilization compared to each other and a sham condition in patients with chronic low back pain: Study protocol for The RELIEF Study. Contemp Clin Trials. 2018 Jul;70:41-52. doi: 10.1016/j.cct.2018.05.012. Epub 2018 May 21. PMID 29792940